CLINICAL TRIAL: NCT04798690
Title: Open, Multi-center, Non-interventional, Prospective/ Retrospective Observational Study on Long-term Safety and Effectiveness of Growtropin®-II Treatment in Children With Short Stature
Brief Title: Long-term Safety and Effectiveness of Growtropin®-II Treatment in Children With Short Stature
Status: Recruiting | Type: Observational
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: DA3002_SS_OS
Record Dates: First submitted 2021-02-17; First posted 2021-03-15 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Growth Hormone Deficiency; Idiopathic Short Stature; Turner Syndrome; Small for Gestational Age
MeSH Terms: conditions — Dwarfism, Pituitary; Turner Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Growth hormone: Growtropin®-II

SUMMARY:
This study evaluates long-term safety and effectiveness of Growtropin®-II treatment in children with short stature.

ELIGIBILITY:
Inclusion Criteria:

* Children with short stature by growth hormone deficiency(GHD) or idiopathic short stature (ISS) or turner's syndrome(TS) or small for gestational age(SGA)
* Children who has official height record at least 6 months prior

Exclusion Criteria:

* Children with Epiphyseal closure

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Short stature by GHD or ISS or TS or SGA
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2021-02-08 (Actual); Primary Completion 2031-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Long term safety assessed through the adverse events | Up to 2 years after epiphyseal closure
  Number of occurrence of treatment-related adverse events

SECONDARY OUTCOMES:
Change of annualized height velocity | Up to 2 years after epiphyseal closure
  To assess the difference in change of annualized height velocity between baseline and every 6 months
The difference between target height and final height | Up to 2 years after epiphyseal closure
  To assess the difference in target height and final height
Changes in Height SDS | Up to 2 years after epiphyseal closure
  To assess the changes in Height SDS between baseline and every 6 months
Changes in skeletal maturity | Up to 2 years after epiphyseal closure
  To assess the changes in skeletal maturity between baseline and every 6 months
Changes in IGF-1 | Up to 2 years after epiphyseal closure
  To assess the changes in IGF-1 between baseline and every 6 months
Changes in IGFBP-3 | Up to 2 years after epiphyseal closure
  To assess the changes in IGFBP-3 between baseline and every 6 months
Changes in BMI SDS | Up to 2 years after epiphyseal closure
  To assess the changes in BMI SDS between baseline and every 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, Seodaemun-gu, South Korea